CLINICAL TRIAL: NCT01615198
Title: A 14 Week, Randomized, Double-blind, Multi-center, Parallel Group, Active Controlled Study to Evaluate the Efficacy and Safety of LCZ696 in Comparison to Olmesartan in Elderly Patients With Essential Hypertension
Brief Title: Efficacy and Safety of LCZ696 in Comparison to Olmesartan in Elderly Patients With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCZ696A2316
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Results first posted 2015-08-18 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Essential Hypertension
Keywords: Hypertension, blood pressure, LCZ696, dual inhibitor, neprilysin, NEP inhibition, vasopeptidase, ARNi, angiotensin receptor
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — olmesartan; sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- LCZ696 (Experimental): Participants were treated with one LCZ696 100 mg tablet and one placebo of LCZ696 every day (qd) for 4 weeks along with placebo of Olmesartan 10 mg capsule qd. Participants were then up-titrated to LCZ 200 mg tablet and one placebo of LCZ696 qd for 6 weeks along with placebo of Olmesartan 20 mg capsule qd. Participants, who did not achieve their goal BP, were uptitrated to 2 LCZ696 200 mg tablets (LCZ696 400 mg) qd for 4 weeks along with placebo of Olmesartan 40 mg capsule qd.
  Interventions: Drug: Placebo; Drug: LCZ696
- Olmesartan (Active Comparator): Participants were treated with olmesartan 10 mg qd for 4 weeks along with 2 placebo of LCZ696 tablets qd. Participants were then uptitrated to olmesartan 20 mg qd for 6 weeks along with 2 placebo of LCZ696 tablets qd. Participants, who did not achieve their goal BP, were uptitrated to olmesartan 40 mg qd for the remaining 4 weeks and 2 placebo LCZ696 tablets qd.
  Interventions: Drug: Olmesartan; Drug: Placebo

INTERVENTIONS:
Drug: Olmesartan — 10 mg, 20 mg, 40 mg capsules
  Arms: Olmesartan
Drug: Placebo — Matching placebo of LCZ696 tablet, matching placebo of Olmesartan capsule
Drug: LCZ696 — 100 mg, 200 mg tablets
  Arms: LCZ696

SUMMARY:
The purpose of this study is to access the efficacy and safety of LCZ696 compared to olmesartan in elderly Asian patients for the treatment of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give written informed consent before any assessment is performed
* Patients with essential hypertension, untreated or currently taking antihypertensive therapy must have a mean sitting systolic blood pressure ≥ 150 mmHg and < 180 mmHg
* Patients must be able to communicate and comply with all study requirements and demonstrate good medication compliance

Exclusion criteria:

* Patients with severe hypertension (msDBP ≥ 110 mmHg and/or msSBP ≥180 mmHg). Patients with history of angioedema, drug-related or otherwise
* Patients with history or evidence of a secondary form of hypertension
* Transient ischemic cerebral attack (TIA) during the 12 months prior to Visit 1 or any history of stroke
* History of myocardial infarction, coronary bypass surgery or any percutaneous coronary intervention (PCI) during the 12 months prior to Visit 1.
* Current angina pectoris requiring medication (other than patients on a stable dose of oral or topical nitrates).
* Patients with Type 1 or Type 2 diabetes mellitus who are not well controlled and are not on a stable dose of antidiabetic medication
* Patients with previous or current diagnosis of heart failure (NYHA Class II-IV).
* Patients with a clinically significant valvular heart disease at the time of screening
* Women of child-bearing potential, who do not use adequate birth control methods Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 588 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (64):
- China (9):
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Hong Kong (3):
  - Novartis Investigative Site, Hong Kong, Hong Kong
  - Novartis Investigative Site, Hong Kong, Shatin, NT
  - Novartis Investigative Site, Hong Kong
- Japan (29):
  - Novartis Investigative Site, Tōon, Ehime
  - Novartis Investigative Site, Chikushi-gun, Fukuoka
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Kyōtanabe, Kyoto
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Toyonaka, Osaka
  - Novartis Investigative Site, Fujimino, Saitama
  - Novartis Investigative Site, Hiki-Gun, Saitama
  - Novartis Investigative Site, Koshigaya, Saitama
  - Novartis Investigative Site, Saitama, Saitama
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Edogawa-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Katsushika-ku, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Kunitachi, Tokyo
  - Novartis Investigative Site, Meguro-ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shibuya-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Tachikawa, Tokyo
  - Novartis Investigative Site, Taitō City, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo
- Philippines (4):
  - Novartis Investigative Site, Quezon City, Manila
  - Novartis Investigative Site, Manila, National Capital Region
  - Novartis Investigative Site, Quezon City
  - Novartis Investigative Site, Valenzuela
- South Korea (10):
  - Novartis Investigative Site, Bucheon-si, Gyeonggi-do
  - Novartis Investigative Site, Goyang-si, Gyeonggi-do
  - Novartis Investigative Site, Seongnam-si, Gyeonggi-do
  - Novartis Investigative Site, Jeonju, Jeollabuk-do
  - Novartis Investigative Site, Koyang, Kyunggi
  - Novartis Investigative Site, Seoul, Seoul
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Daejeon
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
- Taiwan (7):
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LCZ696 | Olmesartan
Started | 296 | 292
Full Analysis Set | 296 | 292
Ambulatory BP Monitoring (ABPM) Subset | 154 | 157
Safety Set | 296 | 292
ABPM Dipper Status Subset | 82 | 84
Completed | 272 | 273
Not Completed | 24 | 19
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Protocol deviation | 1 | 1
Not completed — Physician Decision | 5 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Lack of Efficacy | 1 | 6
Not completed — Adverse Event | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 | Olmesartan | Total
Number analyzed (Participants) | 296 | 292 | 588
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.5 (4.67) | 70.9 (4.67) | 70.7 (4.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 140 | 294
  Male | 142 | 152 | 294

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP)
Description: Sitting BP measurements were performed at trough (immediately prior to dosing at the clinic). At study entry, BP was measured in both arms. The arm with the higher SBP reading was used for the 4 measurements at screening visit and the same arm was used at all subsequent visits. A negative change from baseline indicates improvement.
Time Frame: Baseline, 10 weeks
Population: Only participants, who had both baseline and week 10 values, were included in the analysis. The FAS included all randomized participants who received study medication and had post baseline BP assessments.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 | Olmesartan
Number analyzed (Participants) | 295 | 291
mmHg | -22.71 (0.91) | -16.11 (0.92)

2. Secondary Outcome: Change From Baseline in Mean 24 Hour Ambulatory Systolic Blood Pressure (maSBP)
Description: ABPM over a 24-hour period was conducted at two time-points during the study in a subset of participants. Readings were taken every 20 minutes over the 24 hour period in the non-dominant arm. A negative change from baseline indicates improvement.
Time Frame: Baseline, 10 weeks
Population: A subset of participants, who participated in ambulatory blood pressure monitoring, was analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 | Olmesartan
Number analyzed (Participants) | 154 | 157
mmHg | -14.23 (0.56) | -9.14 (0.56)

3. Secondary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) and Mean Sitting Diastolic Blood Pressure (msDBP)
Description: Sitting BP measurements were performed at trough (immediately prior to dosing at the clinic). At study entry, BP was measured in both arms. The arm with the higher SBP reading was used for the 4 measurements at screening visit and the same arm was used at all subsequent visits. A negative change from baseline indicated improvement.
Time Frame: Baseline, 4 weeks, 14 weeks
Population: Participants from the full analysis set (FAS), who had both baseline and post baseline values at each given time point, were included in the analysis. The FAS included all participants who received study medication and had post baseline BP assessments.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 | Olmesartan
Number analyzed (Participants) | 295 | 291
mmHg
  msSBP, week 4 | -17.64 (0.83) | -15.81 (0.84)
  msDBP, week 4 | -6.08 (0.44) | -5.58 (0.45)
  msSBP, week 14 | -22.53 (0.92) | -16.75 (0.94)
  msDBP, week 14 | -7.92 (0.49) | -5.97 (0.49)

4. Secondary Outcome: Change in Baseline in Mean 24 Hour Ambulatory Diastolic Blood Pressure (maDBP)
Description: as for outcome 2
Time Frame: Baseline, 10 weeks
Population: A subset of participants, who participated in ambulatory blood pressure monitoring, was analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 | Olmesartan
Number analyzed (Participants) | 154 | 157
mmHg | -6.95 (0.31) | -4.47 (0.31)

5. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: Sitting BP measurements was performed at trough (immediately prior to dosing at the clinic). At study entry, BP was measured in both arms. The arm with the higher SBP reading was used for the 4 measurements at screening visit and the same arm was used at all subsequent visits. A negative change from baseline indicates improvement.
Time Frame: Baseline, 10 weeks
Population: Participants from the full analysis set (FAS), who had both baseline and week 10 values, were included in the analysis. The FAS included all participants who received study medication and had post baseline BP assessments.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 | Olmesartan
Number analyzed (Participants) | 295 | 291
mmHg | -8.58 (0.47) | -6.49 (0.48)

6. Secondary Outcome: Change From Baseline in Mean Sitting Pulse Pressure
Description: Pulse rate was with automated BP device after the 4th blood pressure measurement at each visit.
Time Frame: Baseline, 4 weeks, 10 weeks, 14 weeks
Population: Participants from the full analysis set (FAS), who had both baseline and post baseline values at the given time point, were included in the analysis. The FAS included all participants who received study medication and had post baseline BP assessments.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 | Olmesartan
Number analyzed (Participants) | 295 | 291
mmHg
  week 4 | -11.57 (0.60) | -10.38 (0.61)
  week 10 | -14.21 (0.63) | -9.76 (0.64)
  week 14 | -14.65 (0.64) | -10.90 (0.65)

7. Secondary Outcome: Change From Baseline in Daytime and Nighttime maSBP/maDBP
Description: as for outcome 2
Time Frame: Baseline, 10 weeks
Population: A subset of participants, who participated in ambulatory blood pressure monitoring, was analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 | Olmesartan
Number analyzed (Participants) | 154 | 157
mmHg
  maSBP, daytime | -14.32 (0.96) | -10.02 (0.96)
  maSBP, nighttime | -13.97 (0.96) | -7.68 (0.96)
  maDBP, daytime | -7.04 (0.55) | -4.88 (0.56)
  maDBP, nighttime | -6.70 (0.55) | -3.61 (0.56)

8. Secondary Outcome: Change From Baseline in maSBP and maDBP Lowering Based on Nocturnal BP Dipping (Dipper Versus Non-dipper) in Dippers
Description: ABPM over a 24-hour period was conducted at two time-points during the study in a subset of participants. Readings were taken every 20 minutes over the 24 hour period in the non-dominant arm. A non-dipper was defined as a participant who, at baseline, had a mean nighttime ABPM (10 pm - 6 am) that did not drop ≥ 10% below his or her mean daytime ABPM (6 am - 10 pm). A negative change from baseline indicates improvement.
Time Frame: Baseline, 10 weeks
Population: A subset of ABPM participants were considered for the analysis. For each post-dosing hour, only participants with values at baseline and the post dosing hour end point were included in the analysis for that end point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCZ696 | Olmesartan
Number analyzed (Participants) | 82 | 84
mmHg
  maSBP, hour 1 (n=58,66) | -18.48 (14.550) | -14.15 (15.677)
  maSBP, hour 2 (n=62,66) | -20.75 (15.713) | -17.26 (16.843)
  maSBP, hour 3 (n=62,68) | -17.44 (18.884) | -12.65 (18.923)
  maSBP, hour 4 (n=62,68) | -16.90 (16.539) | -14.83 (17.823)
  maSBP, hour 5 (n=61,67) | -16.70 (17.689) | -16.16 (19.460)
  maSBP, hour 6 (n=62,68) | -18.11 (17.856) | -15.00 (19.025)
  maSBP, hour 7 (n=62,68) | -17.60 (18.330) | -14.74 (20.142)
  maSBP, hour 8 (n=62,67) | -15.81 (15.872) | -16.37 (17.552)
  maSBP, hour 9 (n=62,68) | -14.06 (12.877) | -13.55 (19.456)
  maSBP, hour 10 (n=62,68) | -15.55 (15.232) | -13.50 (17.522)
  maSBP, hour 11 (n=62,68) | -13.17 (17.903) | -13.32 (18.198)
  maSBP, hour 12 (n=62,68) | -12.36 (17.222) | -13.43 (20.898)
  maSBP, hour 13 (n=62,68) | -8.71 (19.359) | -10.84 (19.697)
  maSBP, hour 14 (n=62,68) | -7.10 (20.651) | -9.96 (19.663)
  maSBP, hour 15 (n=62,67) | -9.05 (18.528) | -8.68 (17.094)
  maSBP, hour 16 (n=62,68) | -9.90 (17.994) | -7.81 (16.344)
  maSBP, hour 17 (n=62,68) | -9.88 (16.098) | -5.49 (15.031)
  maSBP, hour 18 (n=61,68) | -11.19 (16.482) | -4.88 (13.065)
  maSBP, hour 19 (n=62,68) | -12.38 (15.010) | -6.69 (15.146)
  maSBP, hour 20 (n=62,68) | -15.18 (16.683) | -9.40 (18.217)
  maSBP, hour 21 (n=62,67) | -13.71 (19.977) | -9.04 (15.748)
  maSBP, hour 22 (n=62,68) | -19.28 (19.387) | -9.61 (18.940)
  maSBP, hour 23 (n=60,66) | -16.88 (15.442) | -10.54 (19.470)
  maSBP, hour 24 (n=57,67) | -17.28 (13.472) | -16.03 (19.076)
  maDBP, hour 1 (n=58,66) | -8.34 (9.640) | -7.30 (8.732)
  maDBP, hour 2 (n=62,66) | -9.13 (9.854) | -7.80 (10.747)
  maDBP, hour 3 (n=62,68) | -8.41 (11.698) | -8.21 (9.857)
  maDBP, hour 4 (n=62,68) | -7.35 (10.656) | -8.98 (9.835)
  maDBP, hour 5 (n=61,67) | -8.17 (10.919) | -8.35 (10.282)
  maDBP, hour 6 (n=62,68) | -8.39 (10.623) | -8.09 (12.360)
  maDBP, hour 7 (n=62,68) | -9.14 (11.350) | -7.35 (12.345)
  maDBP, hour 8 (n=62,67) | -7.50 (9.680) | -8.50 (10.839)
  maDBP, hour 9 (n=62,68) | -7.01 (9.374) | -6.65 (12.287)
  maDBP, hour 10 (n=62,68) | -7.83 (9.907) | -6.70 (11.536)
  maDBP, hour 11 (n=62,68) | -8.08 (10.588) | -6.65 (11.023)
  maDBP, hour 12 (n=62,68) | -7.38 (11.993) | -7.64 (13.479)
  maDBP, hour 13 (n=-62,68) | -4.36 (11.325) | -7.16 (12.916)
  maDBP, hour 14 (n=62,68) | -2.70 (13.661) | -6.28 (10.794)
  maDBP, hour 15 (n=62,67) | -4.02 (12.943) | -3.05 (11.417)
  maDBP, hour 16 (n=62,68) | -4.84 (13.097) | -3.88 (10.015)
  maDBP, hour 17 (n=62,68) | -5.71 (12.089) | -3.74 (11.261)
  maDBP, hour 18 (n=61,68) | -5.36 (11.213) | -1.65 (8.939)
  maDBP, hour 19 (n=62,68) | -6.10 (11.197) | -3.42 (9.726)
  maDBP, hour 20 (n=62,68) | -6.75 (10.878) | -4.00 (12.452)
  maDBP, hour 21 (n=62,67) | -6.91 (12.251) | -4.40 (9.746)
  maDBP, hour 22 (n=62,68) | -10.22 (11.394) | -4.48 (11.019)
  maDBP, hour 23 (n=60,66) | -7.85 (9.030) | -5.11 (9.826)
  maDBP, hour 24 (n=57,67) | -7.83 (10.057) | -6.62 (10.418)

9. Secondary Outcome: Change From Baseline in maSBP and maDBP Lowering Based on Nocturnal BP Dipping (Dipper Versus Non-dipper) Status in Non-dippers
Description: as for outcome 8
Time Frame: Baseline, 10 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCZ696 | Olmesartan
Number analyzed (Participants) | 123 | 116
mmHg
  maSBP, hour 1 (n=84,84) | -13.42 (16.050) | -9.53 (18.224)
  maSBP, hour 2 (n=89,85) | -15.60 (18.144) | -8.57 (17.848)
  maSBP, hour 3 (n=90,88) | -13.17 (15.690) | -6.33 (17.694)
  maSBP, hour 4 (n=91,88) | -13.93 (17.260) | -4.98 (16.155)
  maSBP, hour 5 (n=90,88) | -12.90 (19.372) | -4.68 (16.264)
  maSBP, hour 6 (n=90,89) | -12.96 (22.547) | -5.49 (18.843)
  maSBP, hour 7 (n=91,89) | -12.68 (21.126) | -6.64 (17.191)
  maSBP, hour 8 (n=91,88) | -12.65 (18.450) | -7.45 (17.912)
  maSBP, hour 9 (n=91,89) | -13.51 (17.381) | -7.81 (16.968)
  maSBP, hour 10 (n=92,89) | -12.96 (17.350) | -7.63 (18.620)
  maSBP, hour 11 (n=92,89) | -12.69 (18.724) | -6.89 (16.115)
  maSBP, hour 12 (n=92,88) | -13.82 (17.493) | -3.92 (17.244)
  maSBP, hour 13 (n=92,89) | -16.51 (16.485) | -5.49 (18.209)
  maSBP, hour 14 (n=92,88) | -19.39 (16.860) | -5.16 (16.856)
  maSBP, hour 15 (n=92,89) | -19.33 (19.863) | -5.92 (17.627)
  maSBP, hour 16 (n=92,89) | -17.95 (18.731) | -6.57 (18.512)
  maSBP, hour 17 (n=92,89) | -17.34 (17.015) | -12.03 (18.990)
  maSBP, hour 18 (n=92,88) | -16.45 (16.439) | -8.54 (17.397)
  maSBP, hour 19 (n=91,89) | -15.81 (16.349) | -9.33 (17.027)
  maSBP, hour 20 (n=92,89) | -15.33 (15.556) | -6.77 (16.228)
  maSBP, hour 21 (n=91,89) | -14.78 (15.790) | -7.10 (17.961)
  maSBP, hour 22 (n=91,89) | -13.99 (15.653) | -6.05 (15.806)
  maSBP, hour 23 (n=92,85) | -10.93 (14.121) | -8.48 (16.760)
  maSBP, hour 24 (n=86,85) | -14.19 (15.072) | -7.98 (16.160)
  msDBP, hour 1 (n=84,84) | -7.01 (9.033) | -4.59 (10.061)
  msDBP, hour 2 (n=89,85) | -7.39 (10.516) | -3.32 (11.104)
  msDBP, hour 3 (n=90,88) | -6.61 (10.473) | -3.77 (12.284)
  msDBP, hour 4 (n=91,88) | -7.08 (9.826) | -2.24 (11.169)
  msDBP, hour 5 (n=90,88) | -5.75 (13.156) | -1.53 (12.069)
  msDBP, hour 6 (n=90,89) | -7.06 (13.704) | -2.00 (11.418)
  msDBP, hour 7 (n=91,89) | -5.69 (12.453) | -1.70 (11.797)
  msDBP, hour 8 (n=91,88) | -6.13 (10.420) | -3.04 (11.240)
  msDBP, hour 9 (n=91,89) | -7.05 (10.348) | -3.62 (10.743)
  msDBP, hour 10 (n=92,89) | -5.28 (10.221) | -3.14 (10.849)
  msDBP, hour 11 (n=92,89) | -6.18 (11.825) | -3.18 (10.216)
  msDBP, hour 12 (n=92,88) | -6.36 (11.313) | -1.61 (10.970)
  msDBP, hour 13 (n=92,89) | -8.63 (11.364) | -2.41 (10.750)
  msDBP, hour 14 (n=92,88) | -9.68 (11.518) | -1.69 (11.103)
  msDBP, hour 15 (n=92,89) | -9.60 (13.266) | -2.85 (11.012)
  msDBP, hour 16 (n=92,89) | -8.48 (11.992) | -2.54 (11.523)
  msDBP, hour 17 (n=92,89) | -7.60 (9.661) | -5.44 (11.105)
  msDBP, hour 18 (n=92,88) | -8.60 (11.526) | -4.25 (11.062)
  msDBP, hour 19 (n=91,89) | -7.46 (10.284) | -3.93 (11.088)
  msDBP, hour 20 (n=92,89) | -6.21 (10.295) | -3.10 (9.792)
  msDBP, hour 21 (n=91,89) | -7.63 (10.871) | -2.81 (11.002)
  msDBP, hour 22 (n=91,89) | -6.97 (10.589) | -2.60 (10.568)
  msDBP, hour 23 (n=92,85) | -5.72 (9.410) | -2.12 (11.612)
  msDBP, hour 24 (n=86,85) | -6.57 (9.916) | -3.91 (9.240)

10. Secondary Outcome: Number of Participants Achieving Overall Blood Pressure Control in Mean Sitting Systolic Blood Pressure (msSBP) and Mean Sitting Diastolic Blood Pressure (msDBP)
Description: A successful response in overall BP control rate was defined as msSBP < 140 mmHg and msDBP <90 mmHg.
Time Frame: 4 weeks, 10 weeks, 14 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | LCZ696 | Olmesartan
Number analyzed (Participants) | 295 | 291
Participants
  4 weeks | 140 | 120
  10 weeks | 175 | 130
  14 weeks | 173 | 126

11. Secondary Outcome: Number of Participants Achieving Successful Response in msSBP and msDBP
Description: Blood pressure response in msSBP was defined as a mean sitting BP < 140 mmHg or a >=20 mmHg reduction from baseline. Blood pressure response in msDBP was defined as a mean sitting diastolic blood pressure, 90 mmHg or >=10 mmHg reduction from baseline.
Time Frame: 4 weeks,10 weeks, 14 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | LCZ696 | Olmesartan
Number analyzed (Participants) | 295 | 291
Participants
  msSBP, week 4 | 162 | 146
  msSBP, week 10 | 208 | 142
  msSBP, week 14 | 205 | 144
  msDBP, week 4 | 264 | 245
  msDBP, week 10 | 275 | 254
  msDBP, week 14 | 268 | 246

12. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Death
Description: Adverse event monitoring was conducted throughout the study.
Time Frame: 14 weeks
Population: Participants from the safety analysis set were analyzed. The safety analysis set included all randomized participants who received study medication and had post baseline assessments.
Measure: Number; unit: Participants
Arm/Group | LCZ696 | Olmesartan
Number analyzed (Participants) | 296 | 292
Participants
  Adverse events (non-serious and serious) | 141 | 113
  Serious adverse events | 7 | 2
  Deaths | 0 | 0

ADVERSE EVENTS:
Arm/Group | LCZ696 | Olmesartan
Serious Adverse Events (participants affected / at risk) | 7/296 | 2/292
Other Adverse Events (participants affected / at risk) | 49/296 | 44/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=296) | Olmesartan (N=292)
ARRHYTHMIA (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 1
MUSCLE ATROPHY (Musculoskeletal and connective tissue disorders) | 1 | 0
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0
HENOCH-SCHONLEIN PURPURA NEPHRITIS (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=296) | Olmesartan (N=292)
NASOPHARYNGITIS (Infections and infestations) | 24 | 18
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 | 6
HYPERURICAEMIA (Metabolism and nutrition disorders) | 11 | 19
DIZZINESS (Nervous system disorders) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.